CLINICAL TRIAL: NCT03141476
Title: Perioperative Cefuroxime in Obese Patients: Dosage According to the BMI
Brief Title: Adequacy of Perioperative Cefuroxime Dosage According to the BMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. med. Jakob Mueller, Senior Physician, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AntibioticsCefuroximePV5153
Record Dates: First submitted 2017-03-21; First posted 2017-05-05 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Obesity; Drug
Keywords: Surgery; Obesity; Drug; Antibiotics; Cefuroxime
MeSH Terms: conditions — Obesity | interventions — Cefuroxime

STUDY DESIGN:
Intervention Model Description: BMI: <30kg/m*m: 1,5g, 31-50kg/m*m: 3,0g, >50kg/m*m: 4,5g
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cefuroxime 1,5g (Other): BMI <30kg/m*m
  Interventions: Drug: Cefuroxime 1,5g
- Cefuroxime 3g (Other): BMI 30-50kg/m*m
  Interventions: Drug: Cefuroxime 3g
- Cefuroxime 4,5g (Other): BMI >50kg/m*m
  Interventions: Drug: Cefuroxime 4,5g

INTERVENTIONS:
Drug: Cefuroxime 1,5g — Patients with BMI of <30kg/m*m: 1,5 g Cefuroxime
  Arms: Cefuroxime 1,5g
Drug: Cefuroxime 3g — Patients with BMI of 30-50kg/m*m: 3g Cefuroxime
  Arms: Cefuroxime 3g
Drug: Cefuroxime 4,5g — Patients with BMI of >50kg/m*m: 4,5 g Cefuroxime
  Arms: Cefuroxime 4,5g

SUMMARY:
This study evaluates the dosage of perioperative cefuroxime for obese patients. Dosage was increased if the BMI was over 30kg/m*m and as well over 50kg/m*m. Drug levels were measured in blood and tissue.

DETAILED DESCRIPTION:
Cefuroxime is an often used antibiotic for surgery antibiotic prophylaxis to avoid surgical wound infection. In this study the dosage of cefuroxime was adjusted to the BMI:

less than 30kg/m*m: 1,5g 31-50kg/m*m: 3,0g more than 50kg/m*m: 4,5g

Cefuroxime was applicated 30 to 60 minutes before the begin of surgery. Drug Levels in blood and fat tissue were measured at skin cut (30-60 minutes after application of Cefuroxime), 45 minutes after skin cut (75-105 minutes after minutes after application of Cefuroxime) and at the end of surgery (up to 150 minutes after application of Cefuroxime) .

The hypothesis of this study is that adequate drug levels are reached in all groups.

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic Intervention
* BMI < 90 kg/m*m
* age: 18-85 years

Exclusion Criteria:

* known history of allergy to cefuroxime or other cephalosporines
* absent consent skill
* elective open surgery
* preoperative therapy with antibiotics
* patient's denial of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-11-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Serum level of Cefuroxime | 30-60 minutes after application of cefuroxime
  Drug Serum Level at skin cut
Serum level of Cefuroxime | 75-105 minutes after application of cefuroxime
  Drug Serum Level 45 minutes after skin cut
Serum level of Cefuroxime | up to 150 minutes after application of cefuroxime
  Drug Serum Level at the end of surgery
Tissue level of Cefuroxime | 30-60 minutes after application of cefuroxime
  Drug Tissue Level at skin cut
Tissue level of Cefuroxime | 75-105 minutes after application of cefuroxime
  Drug Tissue Level 45 minutes after skin cut
Tissue level of Cefuroxime | up to 150 minutes after application of cefuroxime
  Drug Tissue Level at the end of surgery

SECONDARY OUTCOMES:
Surgical site infections | Time until hospital discharge, estimated time period: up to two weeks
  Incidence of surgical site infections
Hospital Retention period | Time until hospital discharge, estimated time period: 5-7 days
  Length of stay in hospital

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No